CLINICAL TRIAL: NCT01353755
Title: Randomised Double Blind Placebo Controlled Pivotal Study to Evaluate Efficacy and Safety of rPhleum in Adult and Adolescent Patients Suffering From Rhinoconjunctivitis +/- Controlled Asthma
Brief Title: 2nd Pivotal Study rPhleum - Adults and Adolescents With Rhinoconjunctivitis +/-Controlled Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL0906rP; 2009-011504-36 (EudraCT Number)
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Rhinoconjunctivitis; Allergic Asthma
Keywords: specific immunotherapy; SIT

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- recombinant Phleum (rPhleum) allergen cocktail (Experimental): The recombinant Phleum (rPhleum) allergen cocktail is prepared by mixing equivalent volumes of each single allergen adsorbate. The recombinant Phleum (rPhleum) allergen cocktail contains Phleum pratense (Phl p) allergens: Type 1, 2, 5 and 6 at equimolar quatities. The total protein concentration in the highest strength is 200μg protein per 1mL aluminium hydroxide suspension.
  Interventions: Drug: Grass pollen specific immunotherapy
- Placebo (Placebo Comparator): Placebo will be administered in the same way as the test product. Placebo will be identical in terms of appearance to the IMP.
  Interventions: Drug: Placabo

INTERVENTIONS:
Drug: Grass pollen specific immunotherapy — * Strength 1 (0.78μg/mL)
  * Strength 2 (6.25μg/mL)
  * Strength 3 (50μg/mL)
  * Strength 4 (200μg/mL)
  The subcutaneous injections will be administered at intervals of 7 (+ 7 days)during up-titration. For maintenance the injection intervals are prolonged to 4 weeks (+2). The double blind treatment period is 2 years, followed by 1 year open-label treatment for patients previously treated with verum and 3 years open-label treatment for patients previously recieved placebo.
  Arms: recombinant Phleum (rPhleum) allergen cocktail
Drug: Placabo — Placebo will be administered in the same way as the test product. Placebo will be identical in terms of appearance to the IMP.
  Arms: Placebo

SUMMARY:
To evaluate efficacy and tolerability of specific subcutaneous immunotherapy with a cocktail of recombinant major allergens of Timothy Grass Pollen (Phleum pratense) in subjects with rhinoconjunctivitis caused by grass pollen with/without controlled asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Has the subject given informed consent according to local requirements before any trial-related activities?
2. Is the subject a legally competent male or female outpatient?
3. Is the subject aged 12 - 65 year?
4. Does the subject suffer from IgE-mediated seasonal allergic rhinoconjunctivitis with or without asthma (controlled, acc. to GINA 2006) caused by grass pollen documented by

   * skin prick test wheal for grass pollen ≥ 5mm in diameter and
   * histamine (1,0% histamindihydrochloride ) wheal ≥ 3mm and
   * NaCl control reaction < 3mm and
   * EAST result (inhouse Allergopharma) ≥ 1.5kU/L to grass pollens and
   * proven clinical relevance of grass pollen allergy by positive conjunctival provocation testing with grass pollen allergens and
   * main discomfort in the respective months.
   * Does the subject with bronchial asthma at entry have a confirmed diagnosis of asthma and does his asthma has been classified as "controlled" according to GINA guidelines (version 2006) with PEF or FEV1at least 80% of predicted normal?
5. Has the subject been treated with anti-allergic medications for at least 2 years prior to enrolment? (Subjects with perennial and continuously treated asthma have to be excluded, see "exclusion criteria" below.)
6. For female patients: Does the subject use effective contraception and does she have a negative pregnancy test result? (Highly effective methods of birth control are defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectibles, combined or oral contraceptives, some IUDs, sexual abstinence or vasectomised partner. No pharmacological interactions are known for hormonal contraceptives and specific immunotherapeutic preparations.)
7. Does the subject suffer from rhinoconjunctivitis symptoms documented in the subjects diary during the baseline season?
8. Does the subject have demonstrated a symptom-score of at least 4 per day during the week following the peak pollen count in the baseline season?

Exclusion Criteria:

1. Is the subject unable to understand and comply with the requirements of the trial, as judged by the investigator?
2. Is the subject currently participating in any other trial or has the subject participated in any other trial within 30 days before inclusion in this trial?
3. Is/was the subject involved in the planning and conduct of the trial?
4. Is the subject an employee of Allergopharma Joachim Ganzer KG or of one of the trial sites?
5. Is the subject in any relationship of dependence with the sponsor and/or with the investigator?
6. Has the subject been previously enrolled or randomised to treatment in the present trial?
7. Is the subject mentally disabled?
8. Is the subject institutionalised due to an official or judicial order?
9. Does the subject have a positive pregnancy test before the baseline phase?
10. Does the subject use an unacceptable and unreliable contraceptive method during the trial, as judged by the investigator?
11. Is the subject pregnant or within the lactation period?
12. Is the subject seeking to become pregnant?
13. Has the subject undergone previous specific immunotherapy with grass pollen allergens in any formulation?
14. Is the subject currently undergoing any sort of immunotherapy?
15. Has the subject ever undergone specific immunotherapy with unknown allergen or an unsuccessful immunotherapy?
16. For allergens which interfere with the grass pollen season for all participating countries
17. Does the subject suffer from any clinically relevant perennial allergies (e.g. cat, mite) and clinical relevance can not be excluded?
18. Does the subject show a total IgE of > 2000kU/l?
19. Does the subject suffer from clinically relevant rhino-conjunctival or respiratory symptoms related to other reasons?
20. Has the subject a PEF or FEV1 < 80% of predicted normal (ECSC)?
21. Has the subject uncontrolled or partly controlled asthma according to GINA guidelines (version 2006)?
22. Does the subject suffer from perennial and continuously treated asthma?
23. Does the subject suffer from rhinoconjunctival atopy symptoms for 20 years or longer?
24. Does the subject suffer from severe acute or chronic diseases (e.g. Diabetes mellitus type I, malignant neoplasia, chronic renal failure), severe inflammatory diseases (liver, kidneys)?
25. Does the subject suffer from autoimmune diseases, immune-defects including immune-suppression, immune-complex-induced immunopathies?
26. Does the subject suffer from severe psychiatric and psychological disorders including impairment of cooperation (e.g. alcohol or drug abuse)?
27. Does the subject suffer from recurrent seizures?
28. Does the subject suffer from irreversible secondary alterations of the reactive organ (e.g., emphysema, bronchiectasis etc.)?
29. Has the subject any physiological and laboratory variables within/outside normal limits and as reported to be greater than Grade 1 changes according to the FDA Guidance for Industry?
30. Is the subject treated with beta-blockers (locally and systemically)?
31. Has the subject any contraindication for use of adrenalin (e.g., acute or chronic symptomatic coronary heart disease, severe hypertension)?
32. Has the subject completed or has an ongoing treatment with anti-IgEantibody?
33. Has the subject completed or has an ongoing long-term treatment with tranquilizer or other psychoactive drugs?
34. Is the subject treated for allergy or asthma according to severity of symptoms?
35. Is the subject using any prophylactic and any treatment with antiallergic medication in fixed (constant) dosage during the treatment phase of the trial?

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2009-10; Primary Completion 2012-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Rhinoconjunctivitis Symptom-Medication-Score | 2 years
  Change of the AUC of the RC-SMS from the baseline season to the season after 2 years of treatment

SECONDARY OUTCOMES:
adverse events | entire trial
  Safety of treatment during the entire trial period will be assessed by clinical laboratory, vital signs and adverse events displayed by MedDRA SOC and Preferred Term.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Hunzelmann, Prof. Dr., Principal Investigator
Locations (1):
- Allergopharma GmbH & Co. KG, Hamburg, Reinbek, Germany

REFERENCES:
- See also: Click here for information about this trial in the European Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/trial/2009-011504-36/DE